CLINICAL TRIAL: NCT03274674
Title: New Approach to Increasing Gingival Thickness in Individuals With Fine Gingival Phenotype:Injectable Platelet Rich Fibrin (I-PRF)
Brief Title: Use of Injectable-platelet-rich-fibrin (I-PRF) to Thicken Gingival Phenotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: boz002
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Periodontoclasia; Gingiva; Injury; Condition; Blood Clot; Gingiva Disorder
Keywords: PRF; I-PRF; Microneedle; Gingival Thickness; Injectable-Platelet-Rich-Fibrin; Platelet Rich Fibrin
MeSH Terms: conditions — Wounds and Injuries; Disease; Thrombosis; Gingival Diseases | interventions — proliferation regulatory factors, human urine; Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Blinded, Parallel group, Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PRF (Experimental): Venous blood will be taken from the patient every session and I-PRF will be created in the centrifuge.I-PRF injected on one side of bilateral thin gingival thickness.Apply once a week and one month after the end of the injections, the patient will be called to the control.
  Interventions: Other: I-PRF
- I-PRF and Microneedling (Active Comparator): Venous blood will be taken from the patient every session and I-PRF will be created in the centrifuge.Microneedle application plus I-PRF injected on the other side in patients with bilateral region with thin gingival phenotype.Apply once a week and one month after the end of the injections, the patient will be called to the control.
  Interventions: Other: I-PRF

INTERVENTIONS:
Other: I-PRF — Venous blood will be taken from the patient every session and I-PRF will be created in the centrifuge.I-PRF injected on one side of bilateral thin gingival thickness.Microneedle application plus I-PRF injected on the other side in patients with bilateral region with thin gingival phenotype.Apply once a week and one month after the end of the injections, the patient will be called to the control.
  Other Names: I-PRF and Microneedling

SUMMARY:
The main objective of this study is to investigate whether the for individuals with thin gingival thickness who are susceptible to gingival recession, the investigators will use i-PRF with microneedle to increase gingival thickness without the need for surgical procedures

DETAILED DESCRIPTION:
Due to the thin gingival phenotype, gingival recession is a problem. The investigators aimed to increase the gingival thickness using i-PRF with microneedle without considering surgical procedures, considering the positive effects of platelet concentrations on revascularization and wound healing in individuals with bone defect, fenestration and gingival thickness which are prone to gingival recession .

ELIGIBILITY:
Inclusion Criteria:

* Never smokers
* Had no history of systemic disease
* Aged ≥18 years old

Exclusion Criteria:

* Patients with a history of diabetes mellitus or systemic disease
* Patients who were under any medication that was known to influence periodontal tissues
* Patients with hormonal changes such as pregnancy or lactation
* Toothless individuals
* Patients who were clotting disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Gingival thickness (mm) | 2 months
  Change in clinical measures of gingival thickness

SECONDARY OUTCOMES:
Plaque Index (PI) | 2 months
  Change in clinical measures of gingival parameters
Gingival Index (GI) | 2 months
  Change in clinical measures of gingival parameters
Bleeding on probing (BOP) | 2 months
  Change in clinical measures of gingival parameters
Clinical attachment level (CAL) | 2 months
  Change in clinical measures of gingival parameters
Probing pocket depth (PD) | 2 months
  Change in clinical measures of gingival parameters

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Betül Özsağır, Study Chair — Bezmialem VU
Locations (1):
- Zeliha Betül ÖZSAĞIR, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ozsagir ZB, Saglam E, Sen Yilmaz B, Choukroun J, Tunali M. Injectable platelet-rich fibrin and microneedling for gingival augmentation in thin periodontal phenotype: A randomized controlled clinical trial. J Clin Periodontol. 2020 Apr;47(4):489-499. doi: 10.1111/jcpe.13247. Epub 2020 Feb 11. PMID 31912532